CLINICAL TRIAL: NCT04283708
Title: Measuring the Eshetic Difference Between Advancement Genioplasty With and Without Submental Liposuction in Treatment of Skeletal Chin Deficiency in Double Chin Patients
Brief Title: Esthetic Outcome of Isolated Advancement Genioplasty With and Without Submental Liposuction in Treatment of Skeletal Chin Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwan Mohamed Atef Ahmed Lotfy, Marwan Mohamed(marwan.mohamed) principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Omfs337
Record Dates: First submitted 2020-02-14; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Receding Chin
Keywords: Submental liposuction; Advancement genioplasty; Double chin patients
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skeletal chin deficiency (Experimental): Advancement genioplasty with submental liposuction
  Interventions: Procedure: Submental liposuction

INTERVENTIONS:
Procedure: Submental liposuction — Advancement Genioplasty With Submental Liposuction

SUMMARY:
This study is to measure the eshetic outcome of of isolated advancement genioplasty with and without submental liposuction in treatment of skeletal chin deficiency in double chin patients

DETAILED DESCRIPTION:
Many methods used to treat skeletal chin deficiency in double chin patients, the aim of this study is to measure the advancement genioplasty with and without submental liposuction

ELIGIBILITY:
Inclusion Criteria:

* skeletal chin deficiency
* double chin patients
* Ages from 18 to 45
* systemic free

Exclusion Criteria:

* body mass index greater than 28
* ages greater than 45
* systemically diseased

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
% of patient satisfaction | 6 months postoperative
  scale of units/discrets

CONTACTS AND LOCATIONS:
Locations (1):
- Marwan mohamed atef ahmed lotfy, Cairo, Egypt